CLINICAL TRIAL: NCT00671242
Title: Correlation of Angiogenesis With 18F-FMT and 18F-FDG Uptake in Non-Small Cell Lung Cancer
Brief Title: Angiogenesis With Positron Emission Tomography (PET) Tracer Uptake
Acronym: angiogenesis
Status: Completed | Type: Observational
Sponsor: Gunma University (Other)
Collaborators: J~pharma (Industry)
Other Study IDs: kkaira1970
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2008-01

CONDITIONS: Angiogenesis; Non-Small Cell Lung Cancer
Keywords: Fluorine-18-α-methyltyrosine,; Positron emission tomography,; Fluorine-18-fluorodeoxyglucose,; Lung cancer,; Angiogenesis; The median VEGF rate was 45% (range, 10-78%).; High expression was seen in 30 patients (81%, 30/37).; VEGF expression was statistically associated with progressively growing microvessel count.
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- I: L-[3-18F]-α-methyltyrosine (18F-FMT) is an amino-acid tracer for PET. We have conducted a clinicopathologic study to elucidate the correlation of angiogenesis with 18F-FMT and 18F-FDG uptake in the patients with non-small cell lung cancer
- Nuclear

SUMMARY:
Purpose: L-[3-18F]-α-methyltyrosine (18F-FMT) is an amino-acid tracer for PET. We have conducted a clinicopathologic study to elucidate the correlation of angiogenesis with 18F-FMT and 18F-FDG uptake in the patients with non-small cell lung cancer (NSCLC).

Method: Thirty-seven NSCLC patients were enrolled in this study, and a pair of PET study with 18F-FMT and 18F-FDG was performed. Uptake of PET tracers was evaluated with standardized uptake value. VEGF, CD31, CD34, LAT1 and Ki-67 labeling index of the resected tumors were analyzed by immunohistochemical staining, and correlated with the clinicopathologic variables and the uptake of PET tracers.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a thoracotomy within 4 weeks after 18F-FMT PET and 18F-FDG PET study
* Histology is non-small cell lung cancer

Exclusion Criteria:

* Patient who received neoadjuvant chemotherapy or radiotherapy before surgery
* Patients who have insulin-dependent diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Gunma University Graduate School of Medicine, Showa-machi, Maebashi, Gunma, Japan

REFERENCES:
- [Derived] Kaira K, Oriuchi N, Shimizu K, Ishikita T, Higuchi T, Imai H, Yanagitani N, Sunaga N, Hisada T, Ishizuka T, Kanai Y, Endou H, Nakajima T, Endo K, Mori M. Correlation of angiogenesis with 18F-FMT and 18F-FDG uptake in non-small cell lung cancer. Cancer Sci. 2009 Apr;100(4):753-8. doi: 10.1111/j.1349-7006.2008.01077.x. Epub 2009 Jan 12. PMID 19141127